CLINICAL TRIAL: NCT05579691
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose Exploration Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of Subcutaneous CTI-1601 in Adult Subjects With Friedreich's Ataxia
Brief Title: A Double-Blind, Placebo-Controlled, Dose Exploration Study of CTI-1601 in Adult Subjects With Friedreich's Ataxia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Larimar Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN-1601-200
Record Dates: First submitted 2022-10-05; First posted 2022-10-14 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CTI-160l (Experimental): CTI-1601 is a recombinant fusion protein and is intended to deliver human frataxin, the protein deficient in Friedreich's ataxia
  Interventions: Biological: CTI-1601
- Placebo (Placebo Comparator): Placebo Comparator
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: CTI-1601 — CTI-1601 is a recombinant fusion protein and is intended to deliver human frataxin, the protein deficient in Friedreich's ataxia
  Arms: CTI-160l
Other: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of subcutaneous (SC) administration of CTI-1601 over 28 days in subjects with Friedreich's ataxia (FRDA).

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, study evaluating two doses (25 mg and 50 mg) of CTI-1601.

This study will consist of at least 2 cohorts with 12 to 15 subjects participating in each cohort. Subjects will be dosed once daily (QD) for 14 days followed by dosing every other day (QOD) through Day 28.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a genetically confirmed diagnosis of FRDA manifested by homozygous GAA repeat expansions, with repeat sizing (if available) included on the diagnosis report.
2. Subject is biologically male or female, 18 years of age or older at screening.
3. Subject must have a mFARS score ≥ 20 and be able to traverse a distance of 25 feet with or without some assistive device (e.g., cane, walker, crutches, self-propelled wheelchair), and (a) be able to sit upright with thighs together and arms crossed without requiring support on more than two sides; (b) be able to transfer from bed to chair independently or with assistance if, in the opinion of the PI, the degree of physical disability does not result in undue risk to the subject while participating in the study; and (c) perform basic daily care, such as feeding themselves and personal hygiene, with minimal assistance.
4. Subject must weigh > 40.0 kg.

Exclusion Criteria:

Subjects are excluded from the study if any of the following exclusion criteria are met:

1. If the subject previously participated in a study of CTI-1601 (CLIN-1601-101 (NCT04176991) or CLIN-1601-102 (NCT04519567)) the subject may not enroll in this study if they experienced one or more of the following: (a) Serious Adverse Event (SAE) related to study drug; (b) Adverse Event (AE) defined as Grade 3 or higher according to the CTCAE version 5.0 (or higher), related to study drug; (c) some other event that supports the exclusion of the subject from participating in this study as determined by the Sponsor (i.e., an AE considered clinically significant by the Sponsor regardless of whether it met SAE criteria and regardless of CTCAE grade).
2. Subject who is confirmed as compound heterozygous (GAA repeat expansion on only one allele) for FRDA.
3. Subject used an investigational drug or device within 90 days prior to screening.
4. Subject requires use of amiodarone.
5. Subject used erythropoietin, etravirine, or gamma interferon 90 days prior to Screening.
6. Subject use of biotin supplementation that exceeds 30.0 mcg/day, either as part of a multivitamin or as a standalone supplement, within 7 days prior to the first dose of study drug.
7. Subject uses more than 3.0 grams of acetaminophen daily.
8. Subject receives medication that requires SC injection in the abdomen or thigh.
9. Subject received a vaccination within 14 days of administration of the first dose of study drug or is scheduled to receive a vaccination within 14 days after administration of the last dose of study drug. As an exception, influenza and tetanus vaccines must be administered more than 72 hours prior to the first dose of study drug or 72 hours after the administration of the last dose of study drug.
10. Subject has a screening ECHO LVEF < 45%.
11. Male subject has a QTcF > 450 milliseconds or female subject has a QTcF > 470 milliseconds on an ECG.
12. Subject currently receiving or having received omaveloxolone within 30 days prior to Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events | Through study completion, an average of 93 days
  Overall summary of Participants with Treatment Emergent Adverse Events

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of CTI-1601 after multiple doses | At baseline and up to 29 days
  Summary assessment of changes in the maximum observed plasma concentration (Cmax) of CTI-1601 after multiple doses
Area under the concentration time curve (AUC) of CTI-1601 from time 0 through the last measurable time point | At baseline and up to 29 days
  Summary assessment of changes in the AUC of CTI-1601 from time 0 to the last measurable time point and during the dosing interval
Time to maximum observed plasma concentration (tmax) of CTI-1601 after multiple doses | At baseline and up to 29 days
  Summary assessment of the time to maximum observed plasma concentration (tmax) of CTI-1601 after multiple doses
Time to last observed plasma concentration (tlast) of CTI-1601 after multiple doses | At baseline and up to 29 days
  Summary assessment of the time to last observed plasma concentration (tlast) of CTI-1601 after multiple doses
Changes from baseline in frataxin levels in buccal cells | At baseline and up to 58 days
  Summary assessment of changes in frataxin levels in buccal cells
Changes from baseline in frataxin levels in skin punch cells | At baseline and up to 29 days
  Summary assessment of changes in frataxin levels in skin punch cells

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Shenouda, M.D., Principal Investigator — Clinilabs, Inc.
Locations (1):
- Clinilabs Drug Development Corporation, Eatontown, New Jersey, United States

REFERENCES:
- [Background] Delatycki MB, Corben LA. Clinical features of Friedreich ataxia. J Child Neurol. 2012 Sep;27(9):1133-7. doi: 10.1177/0883073812448230. Epub 2012 Jun 29. PMID 22752493
- [Background] Goodkin DE, Hertsgaard D, Seminary J. Upper extremity function in multiple sclerosis: improving assessment sensitivity with box-and-block and nine-hole peg tests. Arch Phys Med Rehabil. 1988 Oct;69(10):850-4. PMID 3178453
- [Background] Koeppen AH. Friedreich's ataxia: pathology, pathogenesis, and molecular genetics. J Neurol Sci. 2011 Apr 15;303(1-2):1-12. doi: 10.1016/j.jns.2011.01.010. PMID 21315377
- [Background] Rudick R, Antel J, Confavreux C, Cutter G, Ellison G, Fischer J, Lublin F, Miller A, Petkau J, Rao S, Reingold S, Syndulko K, Thompson A, Wallenberg J, Weinshenker B, Willoughby E. Clinical outcomes assessment in multiple sclerosis. Ann Neurol. 1996 Sep;40(3):469-79. doi: 10.1002/ana.410400321. PMID 8797541
- [Background] Deutsch EC, Santani AB, Perlman SL, Farmer JM, Stolle CA, Marusich MF, Lynch DR. A rapid, noninvasive immunoassay for frataxin: utility in assessment of Friedreich ataxia. Mol Genet Metab. 2010 Oct-Nov;101(2-3):238-45. doi: 10.1016/j.ymgme.2010.07.001. Epub 2010 Jul 8. PMID 20675166
- [Background] Indelicato E, Nachbauer W, Eigentler A, Amprosi M, Matteucci Gothe R, Giunti P, Mariotti C, Arpa J, Durr A, Klopstock T, Schols L, Giordano I, Burk K, Pandolfo M, Didszdun C, Schulz JB, Boesch S; EFACTS (European Friedreich's Ataxia Consortium for Translational Studies). Onset features and time to diagnosis in Friedreich's Ataxia. Orphanet J Rare Dis. 2020 Aug 3;15(1):198. doi: 10.1186/s13023-020-01475-9. PMID 32746884
- [Background] Lawerman TF, Brandsma R, Burger H, Burgerhof JGM, Sival DA; the Childhood Ataxia and Cerebellar Group of the European Pediatric Neurology Society. Age-related reference values for the pediatric Scale for Assessment and Rating of Ataxia: a multicentre study. Dev Med Child Neurol. 2017 Oct;59(10):1077-1082. doi: 10.1111/dmcn.13507. Epub 2017 Aug 17. PMID 28815574
- [Background] Lazaropoulos M, Dong Y, Clark E, Greeley NR, Seyer LA, Brigatti KW, Christie C, Perlman SL, Wilmot GR, Gomez CM, Mathews KD, Yoon G, Zesiewicz T, Hoyle C, Subramony SH, Brocht AF, Farmer JM, Wilson RB, Deutsch EC, Lynch DR. Frataxin levels in peripheral tissue in Friedreich ataxia. Ann Clin Transl Neurol. 2015 Aug;2(8):831-42. doi: 10.1002/acn3.225. Epub 2015 Jul 1. PMID 26339677
- [Background] Pandolfo M. Friedreich ataxia. Arch Neurol. 2008 Oct;65(10):1296-303. doi: 10.1001/archneur.65.10.1296. PMID 18852343